CLINICAL TRIAL: NCT07233824
Title: Effects of Fun-Core (Child-Friendly Core Stabilization) Exercises on Balance and Functional Mobility in Children With Spastic Cerebral Palsy: A Single-Blind Randomized Controlled Trial
Brief Title: Effects of Fun-Core (Child-Friendly Core Stabilization) Exercises on Balance and Functional Mobility in Children With Spastic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Berk Korkut, Medical Doctor (Res. Assist. Dr.), Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-29624016-050.99-3354321
Record Dates: First submitted 2025-09-29; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hemiplegic Cerebral Palsy; Cerebral Palsy (CP); Core Stabilization; Exercise; Functional Mobility; Balance
Keywords: core stabilization exercises; cerebral palsy; functional mobility; balance; child friendly
MeSH Terms: conditions — Cerebral Palsy; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (G1) (Active Comparator): In addition to a brochure showing the number of sets and repetitions to be given to the patients as a standard home exercise program, the Fun-Core video exercise program, designed as a child-friendly core stabilization exercise program to be performed 3 times a week, will be given to the intervention group (G1), and the exercises will be delivered to the participants through a website with special accounts.
  Interventions: Other: Exercise
- Control Group (G2) (Other): Standard home exercise program (brochure)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Fun-Core Exercises will be narrated, prepared and recorded in video format, and then delivered in order to ensure children's development and motivation.
  Arms: Intervention Group (G1)
Other: Exercise — Standard home based exercise program

SUMMARY:
A total of 54 children, aged between 6 and 12 years, diagnosed with hemiplegic cerebral palsy and not meeting the exclusion criteria, who registered at the outpatient clinics of the Department of Physical Medicine and Rehabilitation, Istanbul University, Istanbul Faculty of Medicine, between June 1, 2025 and March 1, 2026, were planned to be included in our thesis study, which was planned to be prospective, randomized and single-blind. Children and their parents will be informed verbally and in writing about the study's purpose, duration, and method of implementation, and their informed consent will be obtained. They will be asked to sign an "Informed Consent Form." Patient assessment and follow-up forms will be completed at pre- and post-treatment follow-ups. Patients who meet the inclusion criteria will be numbered according to their order of admission and then randomly assigned to either the intervention or control groups by a computer program.

In addition to a brochure showing the number of sets and repetitions to be given to the patients as a standard home exercise program, the Fun-Core video exercise program, designed as a child-friendly core stabilization exercise program to be performed 3 times a week, will be given to the intervention group (G1), and the exercises will be delivered to the participants through a website with special accounts.

The control group (G2) will receive a standard home exercise program in brochure format, showing the number of sets and repetitions. The exercise program will be performed at home three times a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children with hemiplegic cerebral palsy between the ages of 6 and 12
* Children with Gross Motor Function Classification System (GMFCS) Levels 1, 2, and 3
* Shoe sizes 30 and above

Exclusion Criteria:

* Cognitive impairments that prevent understanding and performing simple commands and tasks
* Botulinum toxin injections into the upper and/or lower extremities within the last 6 months
* History of lower extremity or lumbar surgery within the last year
* Presence of uncontrolled severe epileptic seizures
* Presence of severe vision or hearing problems
* Presence of fixed contractures in the lower extremities

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Modified Timed Up & Go Test | Day 1 (before starting treatment), Day 60 (end of treatment), Day 90 (one month after the end of treatment)
  The mTUG test is a modified version of the Timed Up and Go (TUG) test for assessing functional mobility in children. It essentially measures how quickly an individual can perform the skills necessary for daily living activities-sitting, standing, walking, turning, and sitting down again. Unlike the standard TUG test, it includes instructions and environmental conditions tailored to the developmental level and cognitive capacity of children. In our study, the mTUG test will be administered to participants wearing shoes equipped with wearable sensors, and the test duration will be measured through the shoes.
Pediatric Balance Scale | Day 1 (before starting treatment), Day 60 (end of treatment), Day 90 (one month after the end of treatment)
  It will be used to assess balance in children. It consists of 14 items, each item being scored from 0 to 4. The maximum score is 56. The higher the score, the better the child's balance.
  1. sitting to standing
  2. standing to sitting
  3. transfers
  4. standing unsupported
  5. sitting unsupported
  6. standing with eyes closed
  7. standing with feet together
  8. standing with one foot in front
  9. standing on one foot
  10. turning 360 degrees
  11. turning to look behind
  12. retrieving object from floor
  13. placing alternate foot on stool
  14. reaching forward with outstretched arm

SECONDARY OUTCOMES:
Six Minute Walk Test | Day 1 (before starting treatment), Day 60 (end of treatment), Day 90 (one month after the end of treatment)
  It is considered a measurement that assesses an individual's overall functional status. The test assesses the integrated response of respiratory, cardiovascular, skeletal, nervous, and muscular components. A 30-meter track will be used for the test. The total distance walked by the participant over 6 minutes will be recorded in meters. In our study, the 6-minute walk test will be administered to participants wearing shoes equipped with wearable sensors, and the test will be measured through the shoe.
Trunk Endurance Tests | Day 1 (before starting treatment), Day 60 (end of treatment), Day 90 (one month after the end of treatment)
  Performance assessment is conducted by recording the maximum time the individual can maintain the test position. Before each test, the child is asked to maintain the test position for as long as possible. Each test will be repeated three times, and the average time will be recorded. To minimize the risk of injury or psychological distress, the tests will be explained in detail to the children beforehand, and their administration will be demonstrated. Two healthcare professionals will be present during each test to ensure the child maintains proper form and ensure safety.
  Back extension test: Biering-Sørensen position with trunk held horizontal, pelvis/legs strapped; ended at loss of position or 300s.
  Lateral torso test: Full side-bridge with straight body on elbow; stopped when posture broke or 300s.
  Flexor test: Sit-up at 50° support, arms crossed, feet secured; ended when back touched support or 300s.
Pediatric Reach Test | Day 1 (before starting treatment), Day 60 (end of treatment), Day 90 (one month after the end of treatment)
  It is a measurement method that evaluates the dynamic component of balance. The test will be conducted by measuring the distance in centimeters that participants can reach forward, then to the right and left, without lifting their heels while standing upright. The procedures will be explained to participants once, and then they will be asked to perform the exercise three times. They will be expected to hold each position for at least 3 seconds. Measurements where participants lose their balance and lift their feet off the ground will be invalid. The distance reached will be measured in centimeters using a non-stretchable tape measure.
  The test consists of two sections: sitting and standing, with three items in each section (six items in total). The total score is calculated by measuring the distance in centimeters between the starting position (shoulder flexed 90° for forward reach and shoulder abducted 90° for side reach) and the maximum stable reach.
WeeFIM | Day 1 (before starting treatment), Day 60 (end of treatment), Day 90 (one month after the end of treatment)
  The WeeFIM is used to measure functional independence in activities of daily living for children aged 6 months to 12 years. It consists of 18 items covering self-care, toilet control, mobility, locomotion, communication, and social development.
  A 7-level ordinal rating system ranging from 7 (complete independence) to 1 (total assistance), is used to score performance in each item. As with the FIM, the Wee- FIM consists of two dimensions: motor and cognitive.
  The WeeFIM is a reliable and valid tool for assessing the functional status of children with CP.
PEDQoL 4.0 Pediatric Quality of Life Questionnaire | Day 1 (before starting treatment), Day 60 (end of treatment), Day 90 (one month after the end of treatment)
  The PEDQoL 4.0 Pediatric Quality of Life Questionnaire will be used. Depending on the participant's age, the child report and parent report forms will be used for children aged 7 and 8, and the child report and parent report forms for children aged 8-12. It is designed to measure core health dimensions defined by the World Health Organization (WHO). It is administered in parallel in child self-report and parent proxy report formats. The participant is asked how much of a problem each item has been in the past month.
  Participants are asked to rate how problematic each item has been during the past month. Reverse scoring is applied and converted to a 0-100 scale: 0 = 100 points, 1 = 75 points, 2 = 50 points, 3 = 25 points, and 4 = 0 points. The total scale score is calculated by dividing the sum of responses by the number of items answered. If more than 50% of the items are missing, the scale score is not computed.
Children/ Youth with Cerebral Palsy Brief (6-13 years of age) | Day 1 (before starting treatment), Day 60 (end of treatment), Day 90 (one month after the end of treatment)
  Activity and Participation Assessment: Will be evaluated with the Brief ICF Core Set for Children and Adolescents with CP (≥6, <14 Years). Difficulty levels will be evaluated using the ICF Qualifiers. A score of 0 indicates no difficulty (0-4%), 1 mild difficulty (5-24%), 2 moderate difficulty (25-49%), 3 severe difficulty (50-95%), and 4 complete difficulty (96-100%). Scores 8 ("not specified") and 9 ("not applicable") are used when relevant.
  Activity and participation will be assessed under the domains of performance and capacity. Higher scores in each parameter indicate greater limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse R Aydin, MD, Prof., Study Chair — Istanbul University Istanbul Medical Faculty, Department of Physical Medicine and Rehabilitation
Locations (1):
- Istanbul Unıversity, Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Fatih, Turkey (Türkiye)